CLINICAL TRIAL: NCT05117229
Title: Correlation of Spinopelvic Movement With Lateral Radiographs to Assess Spine Motion Prior to Total Hip Arthroplasty
Brief Title: Correlation of Spinopelvic Movement With Lateral Radiographs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Rafael J. Sierra, M.D., Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 21-006428
Record Dates: First submitted 2021-11-01; First posted 2021-11-11 (Actual); Results first posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-10

CONDITIONS: Spinopelvic Relationships as They Relate to Total Hip Arthroplasty's

STUDY DESIGN:
Intervention Model Description: All participants will have the MetaWear Sensors used on them
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- MetaWear Sensor on radiograph (Experimental): subjects being considered for surgical orthopedic surgery will have a MetaWear sensor added to their standard of care lateral sit to stand radiograph
  Interventions: Device: MetaWear Sensor

INTERVENTIONS:
Device: MetaWear Sensor — Sensor placed on the pelvis to record spinopelvic movement. Lateral sitting and standing lumbar radiographs will be taken

SUMMARY:
The purpose of this research is to compare a novel pelvic MetaWear sensor that looks at spine and pelvic movements when taking lateral sit-to-stand radiographs.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide informed consent.
* Hip pathology: 20 presenting for total hip arthroplasty, 20 presenting for joint preservation procedures.

Exclusion Criteria:

- Patients with lumbosacral hardware, contralateral THA, or DJD in the contralateral hip.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-01-19 (Actual); Study Completion 2023-01-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rafael J Sierra, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- MetaWear Sensor on Radiograph: Subjects who had surgical orthopedic surgery had a MetaWear sensor added to their standard of care lateral sit to stand radiograph
  MetaWear Sensor: Sensor was placed on the pelvis to record spinopelvic movement. Lateral sitting and standing lumbar radiographs were taken.
Period: Overall Study
Arm/Group | MetaWear Sensor on Radiograph
Started | 40
Completed | 40
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | MetaWear Sensor on Radiograph
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.6 (18.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 14
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 40
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 31.0 (6.3)

OUTCOME MEASURES:

1. Primary Outcome: Pelvic Tilt (PT)
Description: PT is a position dependent parameter defined as the angle created by a line running from the sacral endplate midpoint to the center of the bifemoral heads and vertical axis. As recorded by theMetaWear sensor reported in degrees.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | MetaWear Sensor on Radiograph
Number analyzed (Participants) | 40
degrees
  Sitting | 40.0 (11.9)
  Standing | 20.0 (10.5)

2. Primary Outcome: Sacral Slope (SS)
Description: Sacral slope (SS) is a position-dependent parameter defined as the angle between a line parallel to the sacral end plate and a horizontal line. As recorded by theMetaWear sensor reported in degrees.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | MetaWear Sensor on Radiograph
Number analyzed (Participants) | 40
degrees
  Sitting | 16.2 (11.0)
  Standing | 33.2 (11.34)

3. Primary Outcome: Pelvic Incidence (PI)
Description: PI is defined as the angle between a line perpendicular to the sacral plate at its midpoint and a line connecting the same point to the center of the bicoxofemoral axis. As recorded by theMetaWear sensor reported in degrees.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | MetaWear Sensor on Radiograph
Number analyzed (Participants) | 40
degrees | 52.0 (12.6)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline to end of study, approximately one day
Arm/Group | MetaWear Sensor on Radiograph
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2021-06-21): https://cdn.clinicaltrials.gov/large-docs/29/NCT05117229/Prot_000.pdf